CLINICAL TRIAL: NCT04786548
Title: A Precision Medicine Approach to OCD Treatment: Targeting Neuroinflammation
Brief Title: Neuroinflammation in Patients With OCD
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: The NYSPI site is currently paused and has been paused since an institutional pause on human subjects research on March 14, 2024.
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Jeffrey Miller, Associate Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 8115
Record Dates: First submitted 2021-03-01; First posted 2021-03-08 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; OCD; Neuroinflammation; Nonsteroidal anti-inflammatory drug; Celecoxib
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Neuroinflammatory Diseases | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Celecoxib Treatment (Experimental): Patients will receive standardized pharmacotherapy with celecoxib 100mg twice daily for the first week, and will then, if well-tolerated, will be increased to 200mg twice daily for the next seven weeks. Visits with the study psychiatrist will occur weekly for the first four weeks, and biweekly thereafter until week 8, which will be conducted remotely in general, although they may be conducted in-person as clinically warranted and may be conducted in person on the days of other in-person visits. If individuals experience significant side-effects from a given dose, the treating physician may lower the medication dose according to clinical judgment; if side-effects are intolerable, we will discontinue the research procedures and advance to open clinical treatment
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib — Patients will receive standardized pharmacotherapy with celecoxib 100mg twice daily for the first week, and will then, if well-tolerated, will be increased to 200mg twice daily for the next seven weeks.
  Other Names: Celebrex

SUMMARY:
The goal of this study is to examine whether measurements of inflammation from brain scanning and blood tests can predict how much benefit patients with obsessive-compulsive disorder (OCD) will have from treatment with an anti-inflammatory medication, celecoxib, when adding to ongoing medication-based treatment for OCD.

DETAILED DESCRIPTION:
Existing evidence-based treatments for adults with obsessive-compulsive disorder (OCD), including cognitive behavioral therapy and first-line medication-based treatment, do not fully resolve symptoms for a majority of patients. This study proposes to test a new treatment strategy for OCD, examining inflammation as one factor that may contribute to the development of OCD and that may be targeted with medication-based treatment. Recent findings using both brain imaging and analyses from blood samples suggest that some individuals with OCD have increased levels of inflammation in the brain, which may have negative effects on brain function, contributing to symptoms of OCD. Moreover, early clinical studies suggest that some medications with anti-inflammatory properties may be beneficial in treating OCD symptoms. An important and untested question is whether the degree of inflammation assessed using these biological tools can predict how much benefit individuals with OCD will derive from treatment with an anti-inflammatory medication. The investigators will measure inflammation in the brain using PET imaging and measures of inflammation in the body using blood tests in adults with OCD. Patients will then undergo 8 weeks of treatment with an anti-inflammatory medication with some evidence of clinical effectiveness in OCD, celecoxib. The investigators predict that OCD patients with greater evidence of inflammation at baseline, assessed by brain imaging and blood tests, will derive the greatest benefit from anti-inflammatory treatment. In addition, the investigators will compare these inflammatory markers with data from a group of healthy volunteers (collected as part of another protocol, IRB #6786), to extend earlier work finding elevated inflammatory markers in adult OCD. Finally, the investigators will examine whether celecoxib treatment in OCD patients results in reductions in measures of inflammation measured from blood samples and whether the degree of anti-inflammatory effect observed biologically is related to improvement in OCD symptoms. The ultimate goal of this line of research is to pave the way for more individually-tailored, effective treatments for adult OCD based on improved understandings of pathological targets, and to validate an anti-inflammatory approach to the treatment of OCD in individuals with evidence of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 55 years old
* Principal diagnosis of Obsessive-Compulsive Disorder (OCD)
* Ongoing OCD symptoms despite current treatment with psychiatric medication
* Capacity to provide informed consent

Exclusion Criteria:

* Psychiatric comorbidities that would increase risk of participation or impact research measures (e.g., suicidality)
* Medical or neurological conditions that would increase risk of participation or impact research measures
* Contraindications to an MRI or PET scan (e.g., metal implants)
* Current use of medications that may interact with study drug or impact research measures (e.g., antipsychotics, corticosteroids, immunosuppressant medications, or daily non-steroidal anti-inflammatory medications)
* Starting a new evidence-based therapy for OCD (e.g., exposure with response prevention) 4 weeks prior to study enrollment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale | Week 8
  The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) is a clinician-administered interview that measures the presence and severity of symptoms of Obsessive-Compulsive Disorder. It consists of 10 questions with scores ranging from 0 to 4, with a possible score ranging from 0 to 40. The primary measure of clinical improvement in this study is the Week 8 YBOCS score. In statistical models, we will co-vary for the Week 0 YBOCS score to account for baseline symptoms severity, but the Week 8 value is the primary outcome.

SECONDARY OUTCOMES:
TSPO Volume of Distribution assessed by PET imaging with [11C]ER-176 | Baseline
  We will perform PET imaging with the [11C]ER-176 radiotracer to quantify TSPO binding, a marker of neuroinflammation, quantified as the outcome measure Volume of Distribution (VT).
MILLIPLEX MAP Human Cytokine/Chemokine Magnetic Bead Panel | Baseline
  This assay from Millipore Sigma simultaneously quantifies 41 cytokine and chemokine biomarkers from serum.
MILLIPLEX MAP Human Cytokine/Chemokine Magnetic Bead Panel | Week 8
  This assay from Millipore Sigma simultaneously quantifies 41 cytokine and chemokine biomarkers from serum.
PGE2 | Baseline
  prostaglandin E2 levels will be measured in serum.
PGE2 | Week 8
  prostaglandin E2 levels will be measured in serum.
PGF2-alpha | Week 0
  Prostaglandin F2-alpha levels will be measured in serum.
PGF2-alpha | Week 8
  Prostaglandin F2-alpha levels will be measured in serum.
CRP | Week 0
  C-reactive protein levels will be measured in serum.
CRP | Week 8
  C-reactive protein levels will be measured in serum.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Miller, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No